CLINICAL TRIAL: NCT06563102
Title: A 12-week, Randomized, Double-Blind, Phase 4 Study Evaluating the Effect of AIRSUPRA Compared to Albuterol Administered as Needed on Changes in Airway Inflammation, Symptoms, and Rescue Therapy Utilization in Adults With Mild Asthma
Brief Title: Study to Investigate Changes in Airway Inflammation, Symptoms, and Rescue Therapy Utilization With AIRSUPRA Compared to Albuterol as Needed in Adults With Mild Asthma
Acronym: DARWIN
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D6930C00018
Record Dates: First submitted 2024-08-19; First posted 2024-08-20 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Mild Asthma
Keywords: Respiratory Hypersensitivity; Asthma
MeSH Terms: conditions — Respiratory Hypersensitivity; Asthma | interventions — Albuterol; Budesonide

STUDY DESIGN:
Intervention Model Description: At Visit 2 (Week 0), participants who demonstrated ≥ 80% compliance with all at-home study procedures during the last 14 days of the Lead-in Period, and who have used their albuterol rescue inhaler at least 2 days per week during the last 14 days of the Lead-in Period (≥ 4 uses total) will be randomized to continue the study and provided with study drug.
  Randomization will be stratified by Visit 1 FeNO level (< 50 ppb / ≥ 50 ppb) and geographic region. Both albuterol/budesonide and albuterol will be supplied in identical inhalers and the maximum daily dose is the same for the 2 IMPs (6 doses, ie, 12 inhalations/day).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both albuterol/budesonide and albuterol will be supplied in identical inhalers and the maximum daily dose is the same for the 2 IMPs (6 doses, ie, 12 inhalations/day).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 - Participants randomized to receive albuterol/budesonide (Experimental): Participants will be randomized based on Visit 1 FeNO levels (< 50 ppb / ≥ 50 ppb) and geographic region. Participants who are randomized to receive albuterol/budesonide for as-needed rescue therapy will be compared to participants randomized to receive albuterol for as-needed rescue therapy.
  Interventions: Combination Product: Albuterol/Budesonide
- Group 2 - Participants randomized to receive albuterol (Active Comparator): Participants will be randomized based on Visit 1 FeNO levels (< 50 ppb / ≥ 50 ppb) and geographic region. Participants who are randomized to receive albuterol/budesonide for as-needed rescue therapy will be compared to participants randomized to receive albuterol for as-needed rescue therapy.
  Interventions: Combination Product: Albuterol

INTERVENTIONS:
Combination Product: Albuterol/Budesonide — Oral Inhalation. Rescue medication. Unit dose strength of 80 μg budesonide and 90 μg albuterol per actuation
  Other Names: AIRSUPRA; BDA MDI HFA
  Arms: Group 1 - Participants randomized to receive albuterol/budesonide
Combination Product: Albuterol — Oral Inhalation. Rescue medication. Unit dose strength of 90μg albuterol per actuation.
  Other Names: AS MDI
  Arms: Group 2 - Participants randomized to receive albuterol

SUMMARY:
The purpose of this study is to compare the efficacy and safety of albuterol/budesonide to albuterol in changes in airway inflammation, asthma symptoms, and rescue therapy utilization in adults with mild asthma.

Study details include:

* The study duration will be up to 15 weeks.
* The treatment duration will be 12 weeks.
* The visit frequency will be once every 4 weeks, with 3 clinic visits and 2 video calls in total.

DETAILED DESCRIPTION:
DARWIN is a randomized, active-comparator, double-blind, parallel-group, Phase IV study evaluating the effect of albuterol/budesonide (AIRSUPRA) compared to albuterol administered as-needed in response to symptoms on changes in airway inflammation, asthma symptoms, and rescue therapy utilization in adults with mild asthma.

Approximately 15 sites in the United States of America will enroll adult participants with mild asthma who use albuterol as a rescue inhaler and who do not take ICS as maintenance therapy.

The study will be divided in 2 periods (Lead-in Period and Treatment Period) and the total duration of the study for each participant could be up to 15 weeks, with a visit frequency of once every 4 weeks:

* Lead-In Period: Up to 3 weeks
* Treatment Period: 12 weeks

ELIGIBILITY:
Inclusion Criteria:

Informed Consent

1 Capable of giving signed informed consent as described in the protocol which included compliance with the requirements and restrictions listed in the ICF and protocol

Type of Participant and Disease Characteristics 3 Diagnosis of asthma, by a prescribing health care professional 4 ≥ 2 prescriptions for a SABA inhaler in the past 12 months prior to Visit 1 (and the expectation that the participant will probably use their rescue inhaler ≥ 2 days per week as this is required at Visit 2 for randomization following the Lead-in Period) 5 FeNO ≥ 25 ppb at Visit 1

Sex and Contraceptive/Barrier Requirements 7 Female participants: Females must be not of childbearing potential or using a form of birth control as defined below:

* Females not of childbearing potential are defined as females who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. The following age-specific requirements apply:

  * Females < 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and in the absence of any alternative medical cause, as judged by the investigator.
  * Females ≥ 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.
* Female participants of childbearing potential must use a highly effective form of birth control. A highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly. Females of childbearing potential who are sexually active with a non-sterilized male partner must agree to use one highly effective method of birth control, as defined below, from enrolment throughout the study and until at least 14 days after last dose of study intervention. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception. Female condom and male condom should not be used together.

  * All females of childbearing potential must have a negative pregnancy test result at Visit 1.
  * Females < 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatment and in the absence of any alternative medical cause, as judged by the investigator.
* Highly effective birth control methods are listed below:

  * Total sexual abstinence is an acceptable method provided it is the usual lifestyle of the participant (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments).
  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:
* Oral
* Intravaginal
* Transdermal

  * Progestogen-only hormonal contraception associated with inhibition of ovulation:
* Oral
* Injectable
* Implantable

  * Intrauterine device or intrauterine hormone-releasing system
  * Bilateral tubal occlusion
  * Male partner sterilization/vasectomy with documentation of azoospermia prior to the female participant's entry into the study, and this male is the sole partner for that participant. The documentation on male sterility can come from the site personnel's review of participant's medical records, medical examination and/or semen analysis or medical history interview provided by her or her partner.

    8 Negative pregnancy test (urine) for female participants of childbearing potential at Visit 1.

Randomization Criteria 5.1.1 at Visit 2 (Week 0)

1. Symptoms requiring rescue medication use for a minimum of 2 days per week for the last 14 days during the Lead-in Period (minimum 4 uses total)
2. At least 80% overall compliance rate for performing daily FeNO and spirometry assessments and completing the twice-daily asthma symptom and rescue medication use diary during the Lead-in Period.

Exclusion Criteria:

Medical Conditions

1. Any significant disease or disorder, or evidence of drug/substance abuse which in the investigator's opinion would pose a risk to participant safety, interfere with the conduct of study, have an impact on the study results, or make it undesirable for the participant to participate in the study.
2. Medical history of life-threatening asthma including intubation and intensive care unit admission.
3. Medical conditions (other than allergic rhinitis) or medications that will influence FeNO, as judged by the investigator.
4. Concurrent respiratory disease: presence of a known pre-existing, clinically important lung condition other than asthma (eg, cystic fibrosis, idiopathic pulmonary fibrosis, pulmonary arterial hypertension, chronic obstructive pulmonary disease).
5. Any disease state or procedure that is likely to necessitate the use of oral/systemic corticosteroids during the Treatment Period, other than asthma.
6. Malignancy: a current malignancy or previous history of cancer in remission for less than 12 months prior to Visit 1 (participants with treated localized squamous cell or basal cell carcinoma of the skin will not be excluded, whereas participants who had melanoma will be excluded). Participants with a history/treatment of malignancy, and which in the investigator's opinion could compromise the safety of the participant.
7. Other concurrent medical conditions: participants who have known, pre-existing, clinically significant cardiovascular (including clinically significant cardiac arrhythmia and participants with known QT interval corrected for heart rate using the Fridericia formula > 480 ms), endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, haematological or any other system abnormalities that are uncontrolled with standard treatment.
8. Current smokers: previous smokers are allowed to be included provided that they stopped smoking > 12 months prior to Visit 1 AND have a smoking history of ≤ 10 pack-years (includes tobacco, e-cigarettes, vapes, marijuana, etc.).
9. Alcohol/substance abuse: a history (or suspected history) of alcohol misuse or substance abuse within 2 years prior to Visit 1.

   Prior/Concomitant Therapy
10. Use of ICS-containing therapy for maintenance or rescue at enrolment. Other therapies for maintenance of asthma control are allowed (leukotriene receptor antagonists and/or antihistamines, for example), but not LAMA or LABA.
11. Use of any systemic or inhaled corticosteroid within 4 weeks of Visit 1
12. Planned use of a nebulizer during the study (between Visits 1 and 5)

    Prior/Concurrent Clinical Study Experience
13. Participation in another clinical study with any marketed or investigational anti-allergic or immunosuppressant biologic drug within 4 months or 5 half-lives (whichever is longer) prior to Visit 1.
14. Participation in another clinical study with a non-biologic investigational product or new formulation of a marketed non-biologic drug during the last 30 days prior to Visit 1.

    Other Exclusions
15. Participants with a known hypersensitivity to the study drugs or any of the excipients of the products.
16. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
17. Previous randomization in the present study.
18. For women only: currently pregnant (confirmed with positive pregnancy test), breastfeeding or planned pregnancy during the study.
19. Planned hospitalization during the study that would interfere with study objectives as judged by the investigator.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to maximum value of daily morning FeNO | Daily over 12 weeks
  Change from baseline to maximum value of daily morning FeNO over 12 weeks of treatment in the albuterol/budesonide group compared to the albuterol group.

SECONDARY OUTCOMES:
Change from baseline in FeNO on high inflammation days | Daily over 12 weeks
  Change from baseline in FeNO on high inflammation days in the albuterol/budesonide group compared to the albuterol group. A high inflammation day is a day in which the FeNO value is ≥ 20 ppb above baseline.
Number of days with high inflammation (annualized rate) | Daily over 12 weeks
  Number of days with high inflammation in the albuterol/budesonide group compared to the albuterol group. A high inflammation day is a day in which the FeNO value is ≥ 20 ppb above baseline.
Number of days with daily morning FeNO measurements ≥ 50 ppb (annualized rate) | Daily over 12 weeks
  Number of days with FeNO >= 50 ppb in the albuterol/budesonide group compared to the albuterol group.
Number of days with daily morning FeNO measurements ≥ 25 ppb (annualized rate) | Daily over 12 weeks
  Number of days with FeNO >= 25 ppb in the albuterol/budesonide group compared to the albuterol group.
Mean absolute difference in daily morning FeNO over 12 weeks of randomized treatment | Daily over 12 weeks
  Mean daily change in FeNO from the median of the individual's daily FeNO measures over 12 weeks in the albuterol/budesonide group compared to the albuterol group.

OTHER OUTCOMES:
Number of SAEs and DAEs | Week 12
  Evaluate the safety and tolerability of albuterol/budesonide compared to albuterol in patients with asthma.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Lancaster, California
  - Research Site, San Diego, California
  - Research Site, Cape Coral, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Plainfield, Indiana
  - Research Site, St Louis, Missouri
  - Research Site, Riverdale, New Jersey
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, North Charleston, South Carolina
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Waco, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPI/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved, AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org